CLINICAL TRIAL: NCT01923714
Title: Impact of a Tolerability Switch to Dorzolamide/Timolol Preservative-free Fixed Combination on Ocular Surface Symptoms in Belgian Glaucoma Patients
Brief Title: Impact of a Tolerability Switch to Dorzolamide/Timolol Preservative-free Fixed Combination on Ocular Surface Symptoms
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S-53534
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2012-12

CONDITIONS: Open Angle Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glaucoma: Patients with open-angle glaucoma (OAG) that require topical intraocular pressure lowering therapy and that were scheduled to switch current therapy to preservative-free DTFC.

SUMMARY:
This study aims at validating in real-life clinical practice and using the self-reported Glaucoma Symptom Scale (GSS) questionnaire, the impact of a switch to preservative-free dorzolamide/timolol fixed combination (DTFC) in patients using preserved topical therapy for glaucoma.

DETAILED DESCRIPTION:
The study is an 8-week multi-center, prospective, observational and non-interventional, open-label study aiming at assessing a change in visual-related quality of life of glaucoma patients that switch therapy to preservative-free DTFC. As a non-interventional study, the decision for the to switch was at the discretion of the physician. Patients scheduled to switch therapy to preservative free DTFC will be asked to fill in the 10 item, linkert-type GSS questionnaire at baseline, at week 4 and at week 8 of therapy switch.

The study data will be collected at a baseline and at 2 follow-up visits occurring 4 weeks +/- 1 week and 8 weeks +/- 1 week. If no visit was scheduled, the patient was asked to send the completed documents to the physician.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients aged over 18 years old at inclusion visit
* Diagnosed as having OAG in one or both eyes
* Who have used the previous preserved eye drops treatment for at least 4 weeks in one eye or both eyes
* Experiencing pre-established ocular surface disease symptoms, as defined in the 2007 report of the International Dry Eye Workshop
* Being scheduled by their ophthalmologist for a switch to preservative-free DTFC eye drops (as monotherapy or replacement of one preserved product of a combined therapy) at inclusion visit due to tolerability issues
* Accepting to participate in the study and who has provided a written informed consent

Exclusion Criteria:

* Patients who had filtering or other ocular surgery within the 6 months preceding the inclusion visit
* Who have already been treated with preservative-free DTFC
* Whose visual acuity is importantly impaired by a severe ocular disease other than OAG, as assessed by the physician
* Currently involved in a clinical trial or study cohort or pharmaco-epidemiology study or interventional study
* With serious mental or physical disability which could interfere with a patient-reported assessment
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with OAG that require topical therapy for intraocular pressure lowering and that were scheduled to switch current therapy to preservative-free DTFC
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in Glaucoma Symptom Scale questionnaire | 8 weeks
  The main study objective was to assess a change in the patient-reported Glaucoma Symptom Scale questionnaire, filled in at baseline (Week 0) and at the end of the 8 week of therapy with preservative-free DTFC.

SECONDARY OUTCOMES:
Change in Functional-related items of the Glaucoma Symptom Scale | 8 weeks
  A secondary outcome was to assess a change in the patient-reported Glaucoma Symptom Scale questionnaire functional parameters, filled in at baseline (Week 0) and week 4 and week 8 of therapy with preservative-free DTFC.
Change in Symptom-related items of the Glaucoma Symptom Scale | 8 weeks
  A secondary outcome was to assess a change in the patient-reported Glaucoma Symptom Scale questionnaire symptomatic parameters, filled in at baseline (Week 0) and week 4 and week 8 of therapy with preservative-free DTFC.

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Stalmans, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Flemish Brabant, Belgium